CLINICAL TRIAL: NCT07243054
Title: Impact of Prepartum Intravenous Fluid Intake on Newborn Weight Loss in the First Days of Life
Acronym: PERLE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2025_843_0037
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Vascular Filling; Newborn; Weight Loss; Jaundice; Respiratory Distress
Keywords: vascular filling; newborn; weight loss; jaundice; respiratory distress
MeSH Terms: conditions — Weight Loss; Jaundice; Dyspnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
At birth, the infant's weight was measured daily to assess the adequacy of nutritional intake. This indicator can be influenced by various factors related to the mother, her pregnancy, as well as medical interventions during the pre-delivery phase, such as pre-partum maternal fluid intakes, and the subsequent feeding method chosen for the newborn infant. This study aimed at exploring the association between maternal vascular fluid loading during labor in the pre-partum period and neonatal weight loss in the first two days of life. The study focuses on infants fedded with infant formula.

This observational, retrospective, single-center study was carried out at the Amiens University Hospital Center. The participants were mothers aged 18 and older, hospitalized in the maternity ward following full-term delivery (> 37 weeks of gestation). Data were collected through the medical records of the patient and their newborn.

The investigators hypothesize that a relationship may exist between maternal pre-partum vascular fluid loading and neonatal weight loss in the first two days of life, in infants fed with infant formula. These results could raise awareness and help adapt medical and parental approaches to neonatal weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Full-term delivery (≥37+0 SA)
* Singleton pregnancy
* Mother over 18 years of age
* Infant formula feeding exclusively in the maternity ward for the first 2 days

Exclusion Criteria:

* Mother under guardianship
* Mother who does not understand French
* Mother objecting to her personal data being reused for research purposes
* Incomplete or incorrectly completed patient medical record
* Mixed or exclusive breastfeeding
* Mother presenting a hemodynamic disorder in the 12 hours preceding delivery, requiring a filling specifically for this reason
* Child with renal pathology or uropathy
* Children with cleft lip, palate or labio-palate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Mother over 18 years of age and newborn
Study Population: Mother over 18 years of age and newborn
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Correlation between maternal vascular fluid loading and newborn infant weight loss | 2 days

SECONDARY OUTCOMES:
Correlation between maternal vascular fluid loading and respiratory distress | 2 days
Correlation between maternal vascular fluid loading and jaundice of the newborn | 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No